CLINICAL TRIAL: NCT00901030
Title: The Association Between Perioperative Platelet Inhibition (Function) and Major Adverse Perioperative Cardiac Events in Post Percutaneous Coronary Intervention Patients Undergoing Non-cardiac Surgery
Brief Title: Association Between Perioperative Platelet Function and Major Adverse Perioperative Events
Status: Completed | Type: Observational
Sponsor: Hamilton Health Sciences Corporation (Other)
Collaborators: University Health Network, Toronto (Other); London Health Sciences Centre (Other); McMaster University (Other)
Responsible Party: Sponsor
Organization: McMaster University (Other)
Other Study IDs: 09-066
Record Dates: First submitted 2009-05-12; First posted 2009-05-13 (Estimated); Last update posted 2015-09-23 (Estimated); Status verified 2015-09

CONDITIONS: Surgery
Keywords: platelet function; perioperative complications; thromboelastography; coronary stents; non-cardiac surgery

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Patients with PCI on blood thinners: Patients have a coronary stent and are taking anti-clotting (anti-platelet) drug and are having non-cardiac surgery.
  Interventions: Procedure: Blood drawn

INTERVENTIONS:
Procedure: Blood drawn — Blood samples will be taken once in the preoperative clinic and once again at the end of the surgery in the post anesthetic care unit to do the TEG and PMA tests.

SUMMARY:
This study will examine the degree of blood thinning (platelet function) in patients coming for non-cardiac surgery on antiplatelet agents using platelet function tests called thromboelastography (TEG) and platelet mapping assay (PMA) and major cardiac complications that occur any time after surgery (perioperative).

DETAILED DESCRIPTION:
Patients who have had stents in their coronary arteries (PCI) have to stay on antiplatelet agents to prevent clotting of their stents. These patients often require non-cardiac surgery (NCS) at some stage after their PCI. The rate of major cardiac complications (MACE)in this population is very high and it is unclear why they are at higher risk than the general population. It is possible their antiplatelet is not adequate, or that surgery causes them to be more clot prone. This is a prospective, multicentre observational study.

ELIGIBILITY:
Inclusion Criteria:

* patients between ages 30-85 years old, receiving post-PCI aspirin and/or clopidogrel therapy
* patients undergoing non-ambulatory, NCS
* patients will have received a bare metal coronary stent within the last 12 months or a drug eluting stent at any time prior to their NCS
* the type of surgery has to be such that there are no contra-indictions to remain on an anti-platelet agent
* surgeon must agree to keep the patient on at least one anti-platelet agent during the perioperative period

Exclusion Criteria:

* clotting abnormalities
* drugs affecting platelet function other than aspirin or clopidogrel
* moderate renal impairment
* liver dysfunction with co-existing thrombocytopenia

Ages: 30 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who have PCI have to stay on antiplatelet agents to prevent clotting of their stents. These patients often require NCS at some stage after their PCI.
Sampling Method: Non-Probability Sample
Enrollment: 250 (Actual)
Dates: Start 2009-03; Primary Completion 2014-10 (Actual); Study Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
Relationship between platelet function and MACE during the perioperative period | 1 month

SECONDARY OUTCOMES:
Association of MACE with perioperative platelet function as measured by TEG and PMA | 1 month

CONTACTS AND LOCATIONS:
Overall Officials: Summer Syed, M.D., Principal Investigator — Hamilton Health Sciences Corporation
Locations (3):
- Canada (3):
  - Hamilton Health Sciences, Hamilton, Ontario
  - London Health Sciences Centre, London, Ontario
  - University Health Network, Toronto, Ontario